CLINICAL TRIAL: NCT01971060
Title: A Case Study to Evaluate Adhesion Risk in Fertility Patients' Post Laparoscopic Myomectomy Utilizing Vloc Suture.
Brief Title: a Study to Evaluate Adhesion Risk in Fertility Patients' Status Post Laparoscopic Myomectomy.
Acronym: VLocmyo
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: The Advanced Gynecologic Surgery Institute (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Charles E Miller MD, President, The Advanced Gynecologic Surgery Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLocmyo
Record Dates: First submitted 2013-09-24; First posted 2013-10-28 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Uterine Fibroids; Infertility
Keywords: uterine fibroids; barbed suture; infertility; adhesions
MeSH Terms: conditions — Leiomyoma; Infertility; Tissue Adhesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- V-Loc suture (Experimental): Laparoscopic surgery utilizing V-Loc suture
  Interventions: Device: surgery utilizing V-Loc suture

INTERVENTIONS:
Device: surgery utilizing V-Loc suture — V-Loc suture will be utilized in the repair of the uterus following removal of fibroid tumors. a second look laparoscopy will be done on all subjects to evaluate scar tissue formation.
  Other Names: Covidien; V-Loc

SUMMARY:
Premenopausal Women ages 18-42 will undergo a laparoscopic myomectomy. Prior to the myomectomy, adhesions will be assessed using a modified AFS scoring technique. All investigators will provide usual and customary care to research subjects during the first look laparoscopy. This includes the use of all standard practice anti-adhesive agents and heparinized irrigation fluids.V-Loc 180 suture will be utilized in all patients. All patients will then be evaluated by means of a second look laparoscopy (SLL) 6-12 weeks after the initial surgery and reevaluated via modified American Fertility Society scoring techniques. An independent reviewer will also score adhesions utilize a video recording made from the second look laparoscopic surgery. Patients will be contacted both 1 and 4 weeks post -op and assessed for complications. It is the expectation that patients will show no greater post-operative adhesion formation and a <1% complication rate. Time and ease of suturing will also be evaluated. It is expected that the V-Loc suturing technique will show significantly reduced suturing time, be easier to use, and will be associated with minimal adhesions.

DETAILED DESCRIPTION:
This is a post-market, controlled, single-center study to evaluate V-Loc suture. 10 subjects will be included in this study. Premenopausal women ages 18-42 will undergo a laparoscopic myomectomy. Adhesion scoring will be done prior to the myomectomy using a modified American Fertility Society scoring technique. V-loc 180 suture will be utilized in all patients for closure of all uterine defects. All patients will then be evaluated by means of a second look laparoscopy (SLL) 6-12 weeks after the initial surgery and evaluated via modified American Fertility Society scoring techniques.

An independent reviewer will also score adhesions utilizing video recordings made from the second look laparoscopic surgery , using the same scoring techniques employed by the PI..

Patients will undergo routine preoperative blood tests in accordance with the Primary Investigators' usual standard of practice. All patients who meet the inclusion criteria will be considered. Patients will be consented prior to entry into the operating room. Surgical time will be measured from start of procedure, start of myomectomy, and start and finish time of each individual uterine closure. All investigators will provide usual and customary care to research subjects during the first look laparoscopy. This includes the use of all standard practice anti-adhesive agents and heparinized irrigation fluids

. Physicians will be surveyed on ease of use and any problems that occur with V-Loc suture.

All patients will be treated with post-operative antibiotics per the Primary Investigator's usual standard of care. Patients will be contacted both one and 4 weeks post surgery and evaluated for complications using a phone survey for pain and bowel functioning. The patient will also have a standard post operative exam with the physician 4-6 weeks post-operatively. A second look laparoscopy will be performed 6-12 weeks following the initial myomectomy. Adhesions will be evaluated using a modified American Fertility Society evaluation tool. Any adhesions seen at the time of SLL will be treated using the physician's preferred method of adhesiolysis. A recording will be obtained of the second look laparoscopy and will be reviewed and scored by an independent reviewer as to the level of adhesions seen .

ELIGIBILITY:
Inclusion Criteria:

Premenopausal female ages 18-42 At least one fibroid 3 cm or greater requiring at least one uterine incision Preparing to undergo Laparoscopic myomectomy

Exclusion Criteria:

Post-menopausal or Pregnant

* Endometriosis involving the uterus
* Adhesions to the uterus found at the time of initial laparoscopy
* History of /Current cancer , except basal cell
* Surgery Contraindications, including cardiac or other major system issue
* Greater than 5 fibroids
* The patient has ever been treated with uterine artery embolization of the myoma or magnetic resonance imaging (MRI) or other guided ultrasonification of myoma(s).
* The patient has any medical condition that might interfere with the safety of surgery and the second look laparoscopy, such as active intra-abdominal infection or abscess
* BMI > 34

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Following Laparoscopic myomectomy utilizing V-Loc 180 suture , Post operative adhesion formation will be measured by an independent reviewer at the time of second look laparoscopy utilizing a scoring tool. | 1 year
  The primary objective of this study is to evaluate post operative adhesion formation after using V-Loc™ 180 during laparoscopic myomectomy.

SECONDARY OUTCOMES:
The time required to close the incision as well as the ease of use to the surgeon will be measured utilizing a 1-5 ease of use scale. | 1 year
  The time required to close the incision as well as the ease of use to the surgeon will be measured .

CONTACTS AND LOCATIONS:
Overall Officials: Charles E Miller, MD, Principal Investigator — Advanced GSI
Locations (1):
- The Advanced gynecologic Surgery Institute, Naperville, Illinois, United States